CLINICAL TRIAL: NCT04440917
Title: Induction Therapy of Camrelizumab Combined With Apatinib Mesylate for Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma (the IMplus Study)
Brief Title: Camrelizumab Combined With Apatinib Mesylate for Head and Neck Squamous Cell Carcinoma
Acronym: IMplus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020HNRT01
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2020-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Inductive therapy with Camrelizumab and Apatinib
  Interventions: Drug: Camrelizumab; Drug: Apatinib Mesylate

INTERVENTIONS:
Drug: Camrelizumab — 200mg, iv, on day 1, 15, 29, 43
  Other Names: Humanized anti-PD-1 inhibitor
Drug: Apatinib Mesylate — 250 mg po, qd, 28 days as a cycle, 2 cycles in total
  Other Names: VEGFR inhibitor

SUMMARY:
This is a prospective, open-labelled study to evaluate the efficacy and safety of camrelizumab combined with apatinib mesylate in the induction treatment of patients with locally advanced head and neck squamous cell carcinoma who were judged surgically unresectable or appropriate for non-surgical definitive therapy. The objective response rate (ORR) and safety will be evaluated as the primary endpoints, the 2-year overall survival (OS) rate and progression free survival (PFS) rate will be the second endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed squamous cell or poorly differentiated or undifferentiated cancer of the head and neck (the primary sites include oral cavity, oropharynx, hypopharynx, larynx, nasal cavity and sinuses);
2. Clinical stage of III-IVb (AJCC 2018);
3. Surgically unresectable and/or refuse surgery or appropriate for non-surgical definitive therapy;
4. Measurable disease;
5. Eastern cooperative oncology group performance status (ECOG PS) score: 0-1;
6. Blood routine: white blood cells> 3,000/mm3, hemoglobin> 8g/L, platelets> 80,000/mm3；Liver function: Alanine Transaminase/Aspartate Transaminase <2.5 times the upper limit of normal, bilirubin <1.5 times the upper limit of normal; Renal function: serum creatinine <1.5 times the upper limit of normal;
7. Sign the informed consent.

Exclusion Criteria:

1. Patients with poor-controlled arterial hypertension (systolic pressure ≥ 140 mmHg and/or diastolic pressure ≥ 90 mm Hg) despite standard medical management;
2. Suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (including QT interval male ≥ 450 ms, female ≥ 470 ms). Grade III-IV cardiac insufficiency according to New York Heart Association (NYHA) criteria or echocardiography check: left ventricular ejection fraction (LVEF)<50%;
3. Has had another active malignancy within the past five years except for cervical cancer in site, in situ carcinoma of the bladder or non-melanoma carcinoma of the skin;
4. Clinically significant and uncontrolled major medical conditions including but not limited to: active uncontrolled infection, symptomatic congestive heart failure, Unstable angina pectoris or cardiac arrhythmia, psychiatric illness/ social situation that would limit compliance with study requirements; any medical condition, which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities;
5. Patients undergoing therapy with other investigational agents;
6. Women who are pregnant or breastfeeding;
7. Patients with any other concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (CR+PR) | 9 weeks
  Objective Response Rate as defined by RECIST 1.1 after induction therapy followed by definitive chemoradiation. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.

SECONDARY OUTCOMES:
Number of Participants With at Least One Grade 3-4 Toxicity | 9 weeks
  Toxicity will be assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4
Overall Survival | 2 years
  Time to death or progression defined by imaging of target lesions via CT or MRI scan every 3 months
Progression-Free Survival | 2 years
  Time to death or progression defined by imaging of target lesions via CT or MRI scan every 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No